CLINICAL TRIAL: NCT07029958
Title: Improved Myeloablative Allogeneic Hematopoietic Stem Cell Transplantation Protocol for the Treatment of Epstein Barr Virus T/NK Lymphoproliferative Disease (EBV-T/NK LPD) and Prevention of Post Transplant Graft-versus-host Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Children's Hospital (Other)
Responsible Party: Principal Investigator, Jun Yang, Doctor, Beijing Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [2024]-Y-254-D
Record Dates: First submitted 2025-06-12; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: EBV-T/NK LPD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental)
  Interventions: Drug: recombinant humanized anti-CD25 monoclonal antibody

INTERVENTIONS:
Drug: recombinant humanized anti-CD25 monoclonal antibody — For children at high risk of GVHD, one of the following conditions must be met (haploidentical donors must meet one condition, while unrelated donors must meet two conditions):
  1. The donor is ≥40 years old;
  2. The donor is an unrelated donor with ≥1 locus mismatch, a haploidentical female donor, or collateral consanguinity (e.g., cousin, uncle/aunt);
  3. Pre-transplant CD3 count ≥4 x 10^8/kg;
  4. The primary disease is in an HLH (hemophagocytic lymphohistiocytosis) flare or active disease phase;
  5. ATG (or biologically equivalent doses of ATLG [1:2] or ALG [1:20]) <10mg/kg. Combining recombinant anti-CD25 humanized monoclonal antibody with conventional pretreatment regimen, before peripheral blood stem cell transfusion (i.e. 0d) and+3d, 1mg/kg，<40kg the maximum dose should not exceed25mg/dose, ≥40kg 1mg/kg, and the maximum dose should not exceed 50mg/dose.

SUMMARY:
To investigate whether the addition of recombinant humanized anti-CD25 monoclonal antibody to the conventional EBV-T/NK LPD conditioning regimen can prevent acute and chronic GVHD after transplantation, improve the severity of GVHD and have a corresponding impact on other related post-transplant complications such as poor engraftment, thrombotic microvascular disease, early EBV reactivation and relapse.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnosis of EBV-T/NK lymphoproliferative disease (EBV-T/NK LPD) according to the ICC2022 diagnostic criteria
* Plan to undergo allogeneic hematopoietic stem cell transplantation (allo HSCT) in our hospital
* Age ≤ 18 years old
* Sign informed consent form
* Meet one of the following conditions (haploid donors must meet one of the above conditions, unrelated donors must meet two of the above conditions): ① donor age≥40 years old; ② The donor source is unrelated donor or haplotype related female or collateral donor (brother sisters, etc.) with ≥ 1 point mismatch; ③ CD3≥4 x 10 ^ 8/kg before transplantation; ④ The primary disease is in an HLH (hemophagocytic lymphohistiocytosis) flare or active disease phase; ⑤ ATG (or ATLG (1:2)/ALG (1:20) equivalent dose)<10mg/kg

Exclusion Criteria:

* The expected survival period for multiple organ failure is no more than 3 months
* Not signing the informed consent form

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2029-10-30 (Estimated); Study Completion 2029-10-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of aGVHD | post-HSCT 100days

SECONDARY OUTCOMES:
Incidence of TMA | post-HSCT 1year
Incidence of VOD | post-HSCT 1year
Overall survival | post-HSCT 1year
Incidence of adverse events | 30 days after discontinuation of medication

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Children's Hospital Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided
The research results will be published in the form of an article in the future. Depending on the circumstances of the study, it may be possible to provide the relevant data upon request via email or other means.